CLINICAL TRIAL: NCT03842787
Title: Role of Anti-ficolin-3 Antibodies in the Pathogenesis of Lupus Nephritis
Brief Title: Anti-ficolin-3 Antibodies in Lupus Nephritis
Acronym: IgFicoLupus
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut de Biologie Structurale Grenoble (Unknown)
Responsible Party: Sponsor
Other Study IDs: 38RC18.303; 2018-A02942-53 (Other: ID RCB)
Record Dates: First submitted 2019-01-22; First posted 2019-02-15 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Systemic Lupus Erythematosus Nephritis
Keywords: systemic lupus erythematosus; lupus nephritis; complement; ficolin-3; anti-ficolin-3 autoantibodies
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SLE patients with lupus Nephritis: 14 SLE patients with lupus Nephritis
  Biological analysis and biopsy were (routinely) performed
  Ethics The protocol will be submitted to a randomly chosen Institutional Review Board (Comité de Protection des Personnes), in compliance to French regulation.
  Investigators will include patients followed for routine care. Patients will be informed that samples (serum and kidney biopsy) that are performed for routine patient care will subsequently be used for research purposes, with no additional blood draw/biopsy. They will sign informed consent.
  Interventions: Other: Biological analysis

INTERVENTIONS:
Other: Biological analysis — Biological and research analysis:
  Quantification of ficolin-3, anti-ficolin-3 antibodies, ficolin-2, anti-ficolin-2 antibodies
  Purification of patients' antibodies (anti-ficolin-3 and -2)
  Evaluation of effects of anti-ficolin-3 and anti-ficolin-2 purified antibodies Investigation of ficolin-3 and ficolin-2 deposition in renal biopsy

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease characterized by the production of multiple autoantibodies and accumulation of immune complexes resulting in systemic inflammatory response and tissue damage. Although the underlying mechanisms are complex, defects in dying cells elimination are likely to contribute to autoantigen overload and development of autoimmunity. Molecules important in damaged cell clearance, such as early complement components, may thus have a protective role. According to this hypothesis, deficiencies in C1q and MBL, the recognition proteins of the classical and lectin pathways of complement; are associated with increased susceptibility to SLE. In the proposed project, the investigators will investigate the involvement of another related recognition protein, ficolin-3, which activates the complement lectin pathway and recognizes necrotic cells. The investigators have shown in a recent study a significant association between the presence of anti-ficolin-3 antibodies and active nephritis in patients with SLE. However, the possible involvement of anti-ficolin-3 antibodies in the pathogenesis of SLE and particularly in lupus nephritis (LN) remains to be elucidated. This project plans to investigate the role of ficolin-3 and ficolin-3 autoantibodies in LN. The study associates two aspects, aiming at deciphering the role of anti-ficolin-3 antibodies in dying cells recognition and investigating the role of ficolin-3 in renal tissue damage. This pilot study will be performed for 14 patients with active LN on serum and renal biopsy, realized for routine patient care. The investigators will explore the effect of anti-ficolin-3 antibodies purified from the patient serum on ficolin-3-dependent necrotic cells recognition, in relation with possible altered clearance of dead cells, which is an important hypothesis of the pathogenesis of SLE. The investigators will also investigate ficolin-3 deposition in renal biopsy, which may contribute to the local formation of immune complexes, leading to complement activation and subsequent inflammation and tissue injury.

DETAILED DESCRIPTION:
PRIMARY OUTCOME MEASURE Exploration of the inhibition of anti-ficolin-3 antibodies purified from the serum of 14 patients with active lupus nephritis in ficolin-3-dependent necrotic cells recognition.

The criterion used is the shift of MFI (Mean Fluorescence Intensity) measured after addition of these antibodies to necrotic Jurkat cells incubated with ficolin-3.

The study has a single visit approach with serum collection, so every outcome is measured at T0, which is the only visit for the patient.

SECONDARY OUTCOME MEASURES

1. Investigation of ficolin-3 deposition in renal biopsy of the same 14 patients with active LN.

   Analysis: deposition of ficolin-3 will be evaluated by immunostaining on renal biopsy.
2. Quantification of anti-ficolin-3 antibodies. Analysis: Anti-ficolin-3 antibodies are quantified by ELISA.
3. Quantification of serum levels of ficolin-3. Analysis: Ficolin-3 is quantified by ELISA.
4. Correlation between anti-ficolin-3 antibodies and serum levels of ficolin-3. Analysis: Anti-ficolin-3 antibodies and ficolin-3 are quantified by ELISA.
5. Correlation between serum levels of anti-ficolin-3 antibodies and ficolin-3 deposition in the kidney.
6. Correlation between serum levels of ficolin-3 and ficolin-3 deposition in the kidney.
7. Exploration of the inhibition of anti-ficolin-2 antibodies purified from the serum of 14 patients with active lupus nephritis in ficolin-2-dependent necrotic cells recognition.

   The criterion used is the shift of MFI (Mean Fluorescence Intensity) measured after addition of these antibodies to necrotic Jurkat cells incubated with ficolin-2.
8. Investigation of ficolin-2 deposition in renal biopsy of the same 14 patients with active LN.

   Analysis: deposition of ficolin-2 will be evaluated by immunostaining on renal biopsy.
9. Quantification of anti-ficolin-2 antibodies. Analysis: Anti-ficolin-2 antibodies are quantified by ELISA.
10. Quantification of serum levels of ficolin-2. Analysis: Ficolin-2 is quantified by ELISA.
11. Correlation between anti-ficolin-2 antibodies and serum levels of ficolin-2. Analysis: Anti-ficolin-2 antibodies and ficolin-2 are quantified by ELISA.
12. Correlation between serum levels of anti-ficolin-2 antibodies and ficolin-2 deposition in the kidney.
13. Correlation between serum levels of ficolin-2 and ficolin-2 deposition in the kidney.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients who have valid health insurance
* Non-opposition to participation obtained
* Diagnostic de lupus according to SLICC 2012, performed more than 3 months ago.
* Active lupus nephritis defined by :

elevated SLEDAI indexes (≥ 4), the presence of a significant proteinuria (≥ 0.5 g/day) and/or the presence of hematuria, aseptic leukocyturia or urinary casts, and documented by renal biopsy and classified according to the ISN/RPS classification.

Non-inclusion Criteria:

* Patient with a known progressing cancer
* Patient who had started lupus nephritis flare treatment
* Participant involved in another interventional clinical study
* Person deprived of liberty by judicial order
* Person under guardianship or curatorship
* Hemoglobin level < 7 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SLE patients with lupus Nephritis
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Exploration of the inhibition of anti-ficolin-3 antibodies purified from the serum of 14 patients with active lupus nephritis in ficolin-3-dependent necrotic cells recognition. | Measure at day of inclusion = TO
  In order to investigate the possible interference of the anti-ficolin-3 antibodies purified from patients'sera with ficolin-3 dependent necrotic cells recognition, recombinant ficolin-3 will be preincubated with the purified specific autoantibodies before addition to Jurkat necrotic cells. Ficolin-3 binding will be measured using the flow cytometry and immunofluorescence assays described above and quantified using the mean fluorescence intensity (MFI). The criterion used is the shift of MFI (Mean Fluorescence Intensity) measured after addition of these antibodies to necrotic Jurkat cells incubated with ficolin-3.

SECONDARY OUTCOMES:
Investigation of ficolin-3 deposition in renal biopsy of the same 14 patients with active LN. | Measure at day of inclusion = TO
  The investigators will investigate the presence of ficolin-3 in the glomeruli by direct immunofluorescence analysis. They search deposits in the interstitial vessels, interstitium and glomeruli (mesangium, extra-membranous, glomerular basement membrane) and quantify them semi-quantitatively (+, ++ or +++).
Quantification of anti-ficolin-3 antibodies. | Measure at day of inclusion = TO
  Anti-ficolin-3 antibodies are quantified by ELISA. Results are given in Arbitrary Units (AU)
Quantification of serum levels of ficolin-3. | Measure at day of inclusion = TO
  Ficolin-3 is quantified by ELISA. Results are given in µg/mL.
Correlation of anti-ficolin-3 antibodies and serum levels of ficolin-3. | Measure at day of inclusion = TO
  Anti-ficolin-3 antibodies and ficolin-3 are quantified by ELISA.
Correlation between serum levels of anti-ficolin-3 antibodies and ficolin-3 deposition in the kidney. | Measure at day of inclusion = TO
  Serum levels of anti-ficolin-3 antibodies and ficolin-3 deposition in the kidney are quantified by ELISA.
Correlation between serum levels of ficolin-3 and ficolin-3 deposition in the kidney. | Measure at day of inclusion = TO
  Serum levels of ficolin-3 and ficolin-3 deposition in the kidney are quantified by ELISA.
Exploration of the inhibition of anti-ficolin-2 antibodies purified from the serum of 14 patients with active lupus nephritis in ficolin-2-dependent necrotic cells recognition. | Measure at day of inclusion = TO
  In order to investigate the possible interference of the anti-ficolin-2 antibodies purified from patients'sera with ficolin-2 dependent necrotic cells recognition, recombinant ficolin-2 will be preincubated with the purified specific autoantibodies before addition to Jurkat necrotic cells. Ficolin-2 binding will be measured using the flow cytometry and immunofluorescence assays described above and quantified using the mean fluorescence intensity (MFI). The criterion used is the shift of MFI (Mean Fluorescence Intensity) measured after addition of these antibodies to necrotic Jurkat cells incubated with ficolin-2.
Investigation of ficolin-2 deposition in renal biopsy of the same 14 patients with active LN. | Measure at day of inclusion = TO
  The investigators will investigate the presence of ficolin-2 in the glomeruli by direct immunofluorescence analysis. They search deposits in the interstitial vessels, interstitium and glomeruli (mesangium, extra-membranous, glomerular basement membrane) and quantify them semi-quantitatively (+, ++ or +++).
Quantification of anti-ficolin-2 antibodies. | Measure at day of inclusion = TO
  Anti-ficolin-2 antibodies are quantified by ELISA. Results are given in arbitrary units (AU).
Quantification of serum levels of ficolin-2. | Measure at day of inclusion = TO
  Ficolin-2 is quantified by ELISA. Results are given in µg/mL.
Correlation between anti-ficolin-2 antibodies and serum levels of ficolin-2. | Measure at day of inclusion = TO
  Anti-ficolin-2 antibodies and ficolin-2 are quantified by ELISA.
Correlation between serum levels of anti-ficolin-2 antibodies and ficolin-2 deposition in the kidney. | Measure at day of inclusion = TO
  Serum levels of anti-ficolin-2 antibodies and ficolin-2 deposition in the kidney are quantified by ELISA.
Correlation between serum levels of ficolin-2 and ficolin-2 deposition in the kidney. | Measure at day of inclusion = TO
  Serum levels of ficolin-2 and ficolin-2 deposition in the kidney are quantified by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- JOUVE, La Tronche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dumestre-Perard C, Clavarino G, Colliard S, Cesbron JY, Thielens NM. Antibodies targeting circulating protective molecules in lupus nephritis: Interest as serological biomarkers. Autoimmun Rev. 2018 Sep;17(9):890-899. doi: 10.1016/j.autrev.2018.03.013. Epub 2018 Jul 29. PMID 30009962
- [Background] Munoz LE, Lauber K, Schiller M, Manfredi AA, Schett G, Voll RE, Herrmann M. [The role of incomplete clearance of apoptotic cells in the etiology and pathogenesis of SLE]. Z Rheumatol. 2010 Mar;69(2):152, 154-6. doi: 10.1007/s00393-009-0603-7. German. PMID 20107814
- [Background] Kravitz MS, Shoenfeld Y. Autoimmunity to protective molecules: is it the perpetuum mobile (vicious cycle) of autoimmune rheumatic diseases? Nat Clin Pract Rheumatol. 2006 Sep;2(9):481-90. doi: 10.1038/ncprheum0290. PMID 16951703
- [Background] Herrmann M, Voll RE, Zoller OM, Hagenhofer M, Ponner BB, Kalden JR. Impaired phagocytosis of apoptotic cell material by monocyte-derived macrophages from patients with systemic lupus erythematosus. Arthritis Rheum. 1998 Jul;41(7):1241-50. doi: 10.1002/1529-0131(199807)41:73.0.CO;2-H. PMID 9663482
- [Background] Honore C, Hummelshoj T, Hansen BE, Madsen HO, Eggleton P, Garred P. The innate immune component ficolin 3 (Hakata antigen) mediates the clearance of late apoptotic cells. Arthritis Rheum. 2007 May;56(5):1598-607. doi: 10.1002/art.22564. PMID 17469142
- [Background] Liphaus BL, Kiss MH. The role of apoptosis proteins and complement components in the etiopathogenesis of systemic lupus erythematosus. Clinics (Sao Paulo). 2010 Mar;65(3):327-33. doi: 10.1590/S1807-59322010000300014. PMID 20360925
- [Background] Sato N, Ohsawa I, Nagamachi S, Ishii M, Kusaba G, Inoshita H, Toki A, Horikoshi S, Ohi H, Matsushita M, Tomino Y. Significance of glomerular activation of the alternative pathway and lectin pathway in lupus nephritis. Lupus. 2011 Nov;20(13):1378-86. doi: 10.1177/0961203311415561. Epub 2011 Sep 5. PMID 21893562
- [Background] Kuraya M, Ming Z, Liu X, Matsushita M, Fujita T. Specific binding of L-ficolin and H-ficolin to apoptotic cells leads to complement activation. Immunobiology. 2005;209(9):689-97. doi: 10.1016/j.imbio.2004.11.001. PMID 15804047
- [Background] Nisihara RM, Magrini F, Mocelin V, Messias-Reason IJ. Deposition of the lectin pathway of complement in renal biopsies of lupus nephritis patients. Hum Immunol. 2013 Aug;74(8):907-10. doi: 10.1016/j.humimm.2013.04.030. Epub 2013 Apr 29. PMID 23639552
- [Background] Tanha N, Pilely K, Faurschou M, Garred P, Jacobsen S. Plasma ficolin levels and risk of nephritis in Danish patients with systemic lupus erythematosus. Clin Rheumatol. 2017 Feb;36(2):335-341. doi: 10.1007/s10067-016-3508-2. Epub 2016 Dec 15. PMID 27981461
- [Background] Colliard S, Jourde-Chiche N, Clavarino G, Sarrot-Reynauld F, Gout E, Deroux A, Fougere M, Bardin N, Bouillet L, Cesbron JY, Thielens NM, Dumestre-Perard C. Autoantibodies Targeting Ficolin-2 in Systemic Lupus Erythematosus Patients With Active Nephritis. Arthritis Care Res (Hoboken). 2018 Aug;70(8):1263-1268. doi: 10.1002/acr.23449. Epub 2018 Jun 21. PMID 29045037
- [Background] Plawecki M, Lheritier E, Clavarino G, Jourde-Chiche N, Ouili S, Paul S, Gout E, Sarrot-Reynauld F, Bardin N, Boelle PY, Chiche L, Bouillet L, Thielens NM, Cesbron JY, Dumestre-Perard C. Association between the Presence of Autoantibodies Targeting Ficolin-3 and Active Nephritis in Patients with Systemic Lupus Erythematosus. PLoS One. 2016 Sep 15;11(9):e0160879. doi: 10.1371/journal.pone.0160879. eCollection 2016. PMID 27631981
- [Background] Trouw LA, Daha MR. Role of anti-C1q autoantibodies in the pathogenesis of lupus nephritis. Expert Opin Biol Ther. 2005 Feb;5(2):243-51. doi: 10.1517/14712598.5.2.243. PMID 15757386